CLINICAL TRIAL: NCT07148453
Title: Effects of Mobile Application-Based Cognitive Training Along With Aerobic Training on Cognitive Impairment and Quality of Life in Stroke
Brief Title: Effects of Mobile Application-Based Cognitive Training Along With Aerobic Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02165/ Umber un Nisa
Record Dates: First submitted 2025-08-24; First posted 2025-08-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; cognitive impairment; Lumosity; brain training games
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumosity-based cognitive training + aerobic exercise (Experimental): The experimental group will receive training through a smartphone-based brain training program using the Lumosity app, as well as aerobic exercise on a bicycle ergometer for 18 sessions other days for 6 weeks, 3 times per week, every session for 40 minutes (20 minutes aerobic training on a stationary bicycle ergometer followed by 20 minutes for Lumosity training application on the smartphone).
  Interventions: Other: Experimental Group
- Aerobics + Traditional mental exercises (Active Comparator): The control group will participate in aerobic training on a bicycle ergometer as well as mental exercises for 18 sessions every other day for 6 weeks, 3 sessions/week, each for 40 minutes.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — The experimental group will receive training through a smartphone-based brain training program using the Lumosity app, as well as aerobic exercise on a bicycle ergometer for 18 sessions other days for 6 weeks, 3 times per week, every session for 40 minutes (20 minutes aerobic training on a stationary bicycle ergometer followed by 20 minutes for Lumosity training application on the smartphone).
  Arms: Lumosity-based cognitive training + aerobic exercise
Other: Control Group — The control group will participate in aerobic training on a bicycle ergometer as well as mental exercises for 18 sessions every other day for 6 weeks, 3 sessions/week, each for 40 minutes
  Arms: Aerobics + Traditional mental exercises

SUMMARY:
This randomized controlled trial will determine the effects of combining mobile application-based cognitive training with aerobic exercise on cognitive function and the effects of combining mobile application-based cognitive training with aerobic exercise on quality of life in post-stroke patients

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines stroke as a clinical syndrome marked by the rapid onset of symptoms indicating a focal or global disturbance in brain function. These symptoms last for more than 24 hours or result in death, with no identifiable cause other than a vascular origin. Data on stroke incidence and prevalence in Pakistan are limited, though numerous case series in the literature highlight notable variations in stroke epidemiology, risk factors, and subtypes within the population. The effects of stroke are vast, encompassing physical disability and mortality as well as profound psychological, social, and economic impacts.

Cognitive ability refers to thinking, making sound decisions, and interacting effectively with one's surroundings. When cognitive ability is impaired, it can affect concentration, memory, and learning. Intelligence, which reflects judgment, understanding, and reasoning skills, is often used to measure cognitive abilities in adapting to the environment. post-stroke cognitive impairment (PSCI) refers to cognitive difficulties that arise within 3 to 6 months after a stroke. These impairments may be linked directly to the stroke site, such as aphasia or memory issues, or result from damage to areas like the hippocampus, thalamus, and certain cortical regions. PSCI often overlaps with vascular cognitive impairment (VCI), displaying challenges in visuospatial, attentional, and executive functions. Although some researchers distinguish between early and delayed PSCI based on the timing of cognitive changes, there is no consistent definition, which has complicated PSCI research.

Mobile brain-training games like Lumosity and Peak aim to enhance cognitive skills, such as working memory and attention, through engaging, gamified tasks. These games use challenges and rewards to boost motivation and support learning. A user of the Lumosity app reported improvements in speed, attention, and memory after consistent use since 2011, with others who have experienced brain injuries such as coma, surgery, or concussion also noting positive effects. Brain-training apps like Lumosity and Peak promote cognitive enhancement through gamified tasks aimed at skills such as memory and attention. These claims have contributed to substantial market growth, with the brain-training app industry projected to exceed USD 44.43 billion by 2030.

Aerobic physical exercise (PE) is potentially significant in alleviating cognitive impairment after a stroke. Several neural mechanisms have been associated with the benefits of aerobic exercise on cognitive recovery. Additionally, aerobic exercise supports angiogenesis, reduces secondary injury, and minimizes neuronal damage, all of which contribute to improved cognitive outcomes following a stroke. Aerobic exercise sessions lasting more than 20 minutes are recommended, depending on the frequency and intensity of the exercise. It is also advisable to include warm-up and cool-down periods of 3 to 5 minutes.

This study evaluates the combined impact of the Lumosity brain-training app and aerobic exercise on cognitive function and quality of life (QoL) in older stroke survivors. Traditional methods typically independently implement cognitive rehabilitation and aerobic training, with limited evidence supporting their combined application. This research aims to demonstrate whether combining these methods yields superior cognitive and functional recovery outcomes. Given the limited research on the use of commercial brain training games specifically for stroke survivors, this study seeks to fill a gap in the literature. Previous research has primarily focused on healthy populations, leaving a need for more targeted investigations in stroke rehabilitation. By assessing Lumosity's impact on cognitive recovery, this study will provide valuable insights into the potential of brain training apps for post-stroke rehabilitation. Furthermore, aerobic exercise has demonstrated significant potential in supporting cognitive recovery after stroke, promoting neural plasticity, enhancing neurogenesis, and improving blood flow to affected brain regions. These mechanisms contribute to better cognitive and functional outcomes. This study will explore the combined benefits of cognitive training and aerobic exercise, investigating whether this integrated approach can offer a more effective, accessible, and low-cost strategy for delaying cognitive decline, improving QoL, and supporting long-term recovery in stroke survivors. If successful, this combined approach could pave the way for scalable, novel interventions that empower stroke survivors in their cognitive rehabilitation and overall recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* Patients aged 30-75 years
* Spasticity grade (1 to 1+) based on the modified Ashworth scale (MAS)
* Patients with CVA Education level: matriculation
* at least Single-event stroke patients,
* with a post-stroke duration of 3 to 18 months.
* Mild to moderate cognitive impairment with a score between 10-25 on MOCA

Exclusion Criteria:

* Patients with a history of recurrent stroke or hemiparesis caused by conditions other than stroke.
* Patients with severe cardiovascular issues (e.g., unstable angina, severe coronary artery disease, or untreated congestive heart failure).
* Patients with dementia, depression, visual or auditory impairments, and other neurological conditions (e.g., Multiple Sclerosis, Parkinson's disease) affecting cognition.
* Individuals on medications known to affect cognitive function.
* Patients with low educational levels (illiterate).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 6 weeks
  Brief cognitive function assessment tool consisting of 12 items. Visuospatial, executive functioning, short-term memory, attention/concentration/Working memory, Language and orientation.
  Normal Cognition= 26-30 Cognitive impairment: Mild=18-25, Moderate=10-17, Severe= under 10
Trail Making Test A and B | 6 weeks
  Measure the cognitive function executive. In part A the patient draws lines to join numbered circles (1-25) to connect them in ascending order. In part B, the patient connects the circles alternating between numbers (1-13) and letters (A-L). Trail A; Average; 29 Sec Deficient; >78 sec Rule of Thumb Most in 90 sec Trail B; Average; 75 sec Deficient; >273 sec. Rule of Thumb Most in 3min
6-Minute Walk Test (6MWT) | 6 weeks
  Submaximal exercise test that assesses aerobic capacity and endurance by measuring the distance an individual can walk on a flat, hard surface in a period of 6 minutes. It reflects functional exercise performance and cardiovascular fitness. Commonly used in stroke rehabilitation to evaluate improvements in mobility and endurance.
Stroke Specific Quality of Life scale (SS-QOL) | 6 weeks
  The self-reported questionnaire consists of 49 items across 12 domains. Mobility, Mood, Self-care, Cognition, Social roles, Upper extremity function, work, sleep, family roles, personality, Vision, and strength. Scoring based on a Likert scale ranging from 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Umber un Nisa, MS-NMPT*, Principal Investigator — Riphah International Unversity
Locations (1):
- Railway General Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No